CLINICAL TRIAL: NCT06099730
Title: Safety and Effectiveness of Pulmonary Vein isOLation And posterioR Wall Ablation wIth pulSed Field Energy in Patients With Paroxysmal and Persistent AF
Acronym: POLARIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Moussa C Mansour, PI, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P002605
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Pulsed Field Ablation (Other): This is a non-randomized one arm study.
  Interventions: Device: Pulsed Field Ablation (PFA)

INTERVENTIONS:
Device: Pulsed Field Ablation (PFA) — PFA using Irreversible Electroporation (IRE) Ablation System

SUMMARY:
The primary objective of this clinical investigation is to demonstrate the safety and 12-month effectiveness of pulmonary vein isolation (PVI) and posterior LA wall isolation in the treatment of subjects with symptomatic paroxysmal and persistent atrial fibrillation using the pulsed field ablation with the VARIPULSE™ catheter and the TRUPULSE™ generator.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal and persistent AF with at least one AF episode electrocardiographically documented within 24 months prior to enrollment. Electrocardiographic documentation may include, but is not limited to ECG, Transtelephonic monitoring (TTM), Zio patch monitor, telemetry strip, or consumer devices
* Age 18-80 years
* Willing and capable of providing written consent
* Able and willing to comply with all pre-, post- and follow-up testing and requirements.

Exclusion Criteria:

* Previous surgical or catheter ablation for AF
* Documented LA thrombus by imaging within 48 hours before procedure (CT, TEE, or intracardiac echocardiogram at the beginning of the procedure).
* Uncontrolled heart failure or New York Heart Association (NYHA) Class IV
* History of blood clotting, bleeding abnormalities or contraindication to anticoagulation (heparin, warfarin, or dabigatran)
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study
* Presence of implanted pacemaker or Implantable Cardioverter-Defibrillator (ICD) or other implanted metal cardiac device that may interfere with the PFA energy field
* Women who are pregnant (as evidenced by pregnancy test if pre- menopausal), lactating, or who are of child-bearing age and plan on becoming pregnant during the course of the clinical investigation
* Life expectancy less than 12 months
* Currently enrolled in an investigational study evaluating another device, biologic, or drug that would interfere with this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of early onset primary adverse events (PAEs) | within seven (7) days of an ablation procedure
Freedom from documented atrial tachyarrhythmia episodes | effectiveness evaluation period (Day 91-Day 365)
Freedom from acute procedural failure | during ablation procedure

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - St. Bernard's Heart and Vascular Center, Jonesboro, Arkansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mount Sinai Hospital, New York, New York
  - Montefiore Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Texas Cardiac Arrhythmia Institute/Research Foundation, Austin, Texas